CLINICAL TRIAL: NCT04901988
Title: Circulating Tumour DNA guidEd Therapy for Stage IIB/C mElanoma After surgiCal resecTION (DETECTION)
Brief Title: Circulating Tumour DNA guidEd Therapy for Stage IIB/C mElanoma After surgiCal resecTION
Acronym: DETECTION
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Closed earlier than expected due to the need for a redesign to reflect the recent change in standard of care guidelines. New design will include these treatments.
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); Manchester Academic Health Science Centre (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp135
Record Dates: First submitted 2021-04-16; First posted 2021-05-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2023-04

CONDITIONS: Melanoma (Skin); Melanoma, Stage II
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Masking Description: No participants were randomised prior to early termination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (No Intervention): In Arm A, patients and clinicians will remain blinded to the ctDNA result and will be managed as per standard of care with regular clinical review and imaging, and treated if they develop evidence of disease recurrence.
- Arm B (Experimental): Patients randomised to Arm B will not be blinded to the positive ctDNA result and will be treated with the intervention.
  Interventions: Drug: Nivolumab 10 MG/ML

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML — Eligible patients randomised to Arm B will receive 480 mg nivolumab monotherapy 4 weekly via IV infusion for up to 2 years.
  Arms: Arm B

SUMMARY:
The trial is looking for new and better ways to treat melanoma, an aggressive type of skin cancer. Having surgery to remove the melanoma will cure the majority of patients with early stage disease. However, a small percentage of these patients will go on to develop further disease, which may spread to other places in their body.

Currently, patients who have been cured of melanoma will have appointments in clinic to check that further disease has not developed or returned and some may also receive regular scans.

The trial team has developed a blood test that tells us whether cancer cells are still present or is becoming active after a patient has been 'cured' of melanoma, even if a scan looks normal. The test looks for pieces of DNA in the blood that are known to have come from the cancer, which we call 'circulating tumour DNA', or ctDNA. Patients who have ctDNA in their blood have an extremely high chance of the cancer returning.

By using the blood test that we have developed we think that we can identify patients earlier than normal. We think that some of the treatments that are used when melanoma cancer has spread may benefit patients at this earlier stage.

We want to see if these patients with ctDNA in their blood, who have a higher risk of their cancer returning or spreading, and receive treatment early have a better response to their cancer compared to those patients who receive treatment when their cancer has returned and it can be seen on a scan. This could mean we would be able to offer patients earlier treatment in the future using just a blood test rather than a scan, while also providing reassurance to those patients that do not have ctDNA in their blood that they do not need treatment and their cancer is not returning.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
3. Histological confirmation of cutaneous melanoma
4. ≥ 18 years.
5. Stage IIB or IIC melanoma (sentinel lymph node (SNLB) staged) according to AJCC version 8 (4).
6. Complete resection (including SNLB) must have been performed within 12 weeks prior to registration.
7. Disease-free status documented both clinically and radiologically within 4 weeks prior to registration.
8. Mutation confirmed in at least one of the following BRAF (p.V600E/p.V600K/p.V600R) /NRAS (p.Q61R/p.Q61K, p.Q61L/p.G12D), which can be tracked in ctDNA with exact point mutation known.
9. ECOG performance status 0/1.
10. Adequate organ function and screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Absolute neutrophil count (ANC) ≥1.5x109/L, Platelets ≥100 x109/L, Haemoglobin ≥90 g/L, Creatinine ≤1.5x ULN or creatinine clearance >30mL/minute using Cockcroft-Gault, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 x ULN unless the patient has familial hyperbilirubinaemia.
11. LDH ≤1.5x ULN as per local institution parameters.
12. Patients who are pregnant or breastfeeding will be eligible to join the trial. However, if they are allocated to Arm B, women of childbearing potential (WOCBP) must agree to have a serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) and must be withdrawn if pregnant or breastfeeding. WOCBP and males who are sexually active with WOCBP must also agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 months for WOCBP or plus 7 months for males who are sexually active with WOCBP (if randomised to Arm B or while receiving any systemic treatment and to follow local guidance if given on Arm A). See Appendix A for further information.

Exclusion Criteria:

1. If previously received prior immunotherapy, chemotherapy, cancer directed vaccine therapy or BRAF/MEK targeted therapy for cancer.
2. Patients with active, known or suspected autoimmune disease. Patients with type 1 diabetes mellitus, rheumatoid arthritis not requiring disease modifying drugs, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger will be permitted to enrol.
3. Current other malignancy or history of another malignancy within the last 3 years. Patients who have been disease-free for 3 years, (i.e. patients with second malignancies that have been definitively treated at least 3 years ago) or patients with a history of completely resected non-melanoma skin cancer are eligible.
4. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the patient's safety, obtaining informed consent, or compliance with study procedures.
5. Patients with a condition requiring ongoing/long-term (>3 months) systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications. Inhaled or topical steroids and adrenal replacement steroid doses ≤10 mg daily prednisolone equivalent are permitted in the absence of active autoimmune disease.
6. Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
7. History of allergies or adverse drug reaction to any of the study drug components or to any monoclonal antibody.
8. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
9. Prisoners or patients who are involuntarily incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomisation until death by any cause, assessed up to 84 months.

SECONDARY OUTCOMES:
Relapse Free Survival | From randomisation to radiological (recist v1.1)/clinical (confirmed histologically) progression, assessed up to 84 months.
Distant metastasis free survival(DMFS) | From randomisation to distant metastatic relapse or death, assessed up to 84 months.
Progression-free survival (PFS) on first line therapy (commenced in Arm A at relapse, and Arm B from randomisation). | From start of treatment (day of first dose) until disease progression defined as clinical (confirmed pathologically) or radiological (recist v1.1) progression or death, assessed up to 84 months.
Time from randomisation to disease progression on first line systemic therapy (Arm A first systemic therapy given at relapse, and Arm B nivolumab from randomisation). | Time from randomisation to disease progression on first line systemic therapy (Arm A first systemic therapy given at relapse, and Arm B nivolumab from randomisation), assessed up to 84 months.
Radiological response in Arm A (CR, PR, SD and PD) and PD vs. no PD in Arm B to first line systemic therapy. | Radiological response in Arm A (CR, PR, SD and PD) and PD vs. no PD in Arm B to first line systemic therapy, assessed up to 84 months.
Time from registration to ctDNA detection. | Time from registration to ctDNA detection, assessed at registration and then every 3 months (year 1 to 3) and every 6 months (year 4 and 5).
Number of patients with undetectable ctDNA (not detectable according to the DETECTION assay), but clinical/radiological progression and site of progression (local or distant in addition to organ site). | From registration to clinical/radiological progression with undetectable ctDNA, assessed up to 84 months.
RFS of patients with undetectable ctDNA (not randomised) vs. patients with detectable ctDNA in Arm A. | From registration to radiological (recist v1.1)/clinical (confirmed histologically) progression in not randomised and in Arm A participants, assessed up to 84 months.
DMFS of patients with undetectable ctDNA (not randomised) vs. patients with detectable ctDNA in Arm A. | From registration to distant metastatic relapse or death in not randomised and in Arm A participants, assessed up to 84 months.
OS defined as time from registration until death of patients with undetectable ctDNA (not randomised) vs. patients in Arm A. | From registration until death of patients with undetectable ctDNA (not randomised) vs. patients in Arm A, assessed up to 84 months.
To assess treatment-free survival. | Time to first line therapy cessation, assessed up to 84 months.
  Defined as the area between Kaplan-Meier curves between time to first line therapy cessation defined as time from initiation of first line therapy until its cessation and time to subsequent therapy initiation or death defined as time from initiation of first line therapy until initiation of subsequent systemic anticancer therapy or death in Arm A vs. Arm B.
Toxicity measured according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | From consent until the end of the trial or until disease progression and at least 100 days post the last treatment dose of nivolumab, assessed up to 84 months.
Health economics assessment as assessed by EQ-5D-5L and resource use questionnaires. | At registration and every 6 months for both monitoring and post randomisation, with an additional questionnaire at baseline prior to therapy on Arm B and at relapse and every 6 Mo until relapse on first line therapy on Arm A, assessed up to 84 months.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lorigan, Professor, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the trial, after the primary results have been published, the de-identified individual participant data (IPD) and associated documentation (e.g. protocol, statistical analysis plan, annotated blank CRF) will be prepared in order to be shared with external researchers. All requests for access to the IPD will be reviewed by an internal committee at the Clinical Trials Unit (CTU) and discussed with the Chief Investigator in accordance with the CTU policy on data sharing. All data sharing must be authorised by the Sponsor.
Time Frame: Early termination of the study was declared prior to any patients being randomised which means we are unable to perform any evaluation of result or outcome.

REFERENCES:
- See also: HRA summary of results- there are no study results due to early termination. See HRA summary link for more details. — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/detection-2/